| Official Title: | Expanding Clinical Trial Awareness among Black |
|-----------------|------------------------------------------------|
| | Communities through Digital Engagement |
| NCT Number: | NCT06218615 |
| Document Type: | Informed Consent Form |
| Date of the | 11/16/23 |
| Document: | |

#### Fred Hutchinson Cancer Center

#### Consent to take part in a research study:

# Expanding Clinical Trial Awareness among Black Communities through Digital Engagement

*Principal Investigator*: Vida Henderson PhD, Fred Hutchinson Cancer Center [206-667-6355]

#### Important things to know about this study.

You are invited to participate in a research study. The purpose of this research is to learn more about the ability of a public service announcement video, developed with input from Black community members, to support awareness and decision making about clinical trial particiation in Black individuals who currently or have ever had a cancer diagnosis.

People who agree to participate in this study will be asked to complete an online survey. You will first be asked a few questions to determine if you are eligible to participate in the study. If you are eligible to participate in the study, you will be asked to answer a short survey about your opinions and beliefs about clinical trials. After that you will watch a short 2- minute video about clinical trials, then answer a few more questions. The study will take about 15 minutes to complete.

You do not have to join this study. Although the study will not benefit participants directly, we hope the information we learn will help increase awareness of and participation in clinical trials among Black individuals in the future.

Following is a more complete description of this study. Please read this description carefully. It is your choice whether or not you decide to participate in this study. At the end of this description, you will be able to choose yes to indicate your consent to participate in the study or you can choose no to decline participation. If you choose to participate, you will automatically be forwarded to the study survey questions.

#### We would like you to join this research study.

We are doing a research study to examine the impact of a culturally tailored video on views and attitudes related to cancer clinical trials.

Since you are an individual who identifies as Black/African American and are 18 years of age or older, and are currently or were prior diagnosed with cancer, we would like to ask you to join this study. We will enroll up to 100 people. Although the study will not benefit participants directly, we hope the information we learn will help increase awareness about clinical trials.

If you agree to be in this study, you will answer a few questions to determine if you are able to participate in the study. If you are eligible to participate in the study, you will be asked to answer questions about yourself and about your opinions and beliefs about the healthcare system and clinical trials. After that you will watch a 2-min educational video (PSA) about clinical trials. You will then answer a few more questions about your opinions and beliefs. The questionnaire including the educational video takes about 15 minutes to complete.

You do not have to be in this study. You are free to say yes or no, or to drop out after joining. There is no penalty or loss of benefits for saying no or dropping out. If you leave the study, your test results and information cannot be removed from the study records.

# Protecting your Privacy as an Individual and the Confidentiality of Your Personal Information

Some organizations may need to look at your survey data for quality assurance or data analysis. These include:

- Researchers involved with this study.
- Fred Hutchinson Cancer Center.
- Institutional Review Boards (IRB), including the Fred Hutchinson Cancer Center IRB. An IRB is a group that reviews the study to protect your rights as a research participant.

We will assign a random number to your survey. The researchers will not have access to your name or other personal information. They will know the random number only. Thus the risk of someone connecting any study information with you as an individual is unlikely.

We will keep your personal information confidential. But we cannot guarantee total confidentiality. Your personal information may be disclosed if required by law.

We will not use your personal information in any reports about this study, such as journal articles or presentations at scientific meetings.

#### Will you pay me to be in this study?

If you **complete** this study, you will be paid \$66 by Qualtrics.

#### How much will this study cost me?

There are no costs for being in this study.

#### What are the main risks of the study?

There are no physical or emotional risks to this study. The main potential risks are a loss of privacy and confidenality, however only Qualtrics will have access to identifying information. No individuals will be identified in any reports from the study. No information will be released that could lead to identification of any participating individual.

#### Do I have to participate in the whole study?

Participating in this study is completely voluntary. You may stop the survey at any time, or choose not to answer some questions.

#### Will my information ever be use for future research?

Your information will not be used for any research other than this study.

### Questions about the study?

If you have questions or complaints about this study, please call Dr. Henderson at 206-667-6355 or email at vahender@fredhutch.org. If you have questions about your rights as a research participant, call the Director of the Fred Hutch Institutional Review Office at 206-667-5900 or email irodirector@fredhutch.org.

## **Signatures**

Please select "I agree" below if you:

- have read this form (or had it read to you); and
- agree to participate in this study.

By selecting "I agree" you are consenting to the conditions described above

- o I agree
- o I disagree